CLINICAL TRIAL: NCT07218640
Title: Aimmune Therapeutics Manufacturing, LLC Longitudinal Collaboration Study: Evaluating the Impact of Lifestyle Factors on the Microbiome
Brief Title: Aimmune Longitudinal Collaboration Study
Acronym: FIBER-IMPACT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aimmune Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: MSRD001
Record Dates: First submitted 2025-10-15; First posted 2025-10-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Stool Spore Colony Forming Units; Microbiome Composition; Dietary Fiber; Stress
Keywords: Spore Colony-Forming Units; Dietary fiber; Stress; Microbiome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baseline Diet (No Intervention): Participants will consume their baseline diet for 8 weeks
- Chia seeds daily (Experimental): Participants will consume 2.5 tbsp chia seeds daily for 8 weeks
  Interventions: Other: Chia seeds

INTERVENTIONS:
Other: Chia seeds — Participant will add 2.5 tbsp daily chia seeds to their diet for 8 weeks
  Arms: Chia seeds daily

SUMMARY:
This study will include healthy households around the Irvine, CA area (based local to employees) and Tempe, AZ and Philadelphia, PA sites that will be instructed to take a daily fiber supplement (2.5 tablespoons of chia seeds [~10.3g of fiber] which is one serving) for two months. Participants will use a stool sampling tool to facilitate ease of stool collection, or they may donate at a study site. Half of participants will add chia seeds to their diet at the beginning of the study and then return to their baseline diet for the second half of the study; half of participants maintain their baseline diet for the first half of the study and add chia seeds to their diet at the second half of the study as a cross-over design. Households (or individual participants, if their household is not participating) will be chosen at random to decide who implements the intervention in the first half versus the second half of the study. Data measurement including metabolomics and sequencing of stool samples, blood sampling for biobanking, stool IgA analysis, stress and diet evaluations will occur initially and throughout the study. Lifestyle questionnaires including but not limited to diet surveys, stress, or depression screening may be collected through electronic forms or telephonically. During enrollment, participants may be asked to complete questionnaires focused on medical, family, dietary, and social histories.

At the end of the study, donor microbiota samples from individuals that are IgA low (undetectable) throughout the study will be evaluated from the presence of microbes that can degrade IgA. If investigators find this is the case, investigators will screen for microbes that can degrade IgA. For individuals that show persistent high fecal IgA or show a substantial improvement in IgA, investigators will transplant fecal samples or spores from fecal samples into germ-free mice to further understand the microbiome and pathophysiology relationship. For the latter, the investigator's hypothesis is that fiber exposure of a specific type will reprogram the microbiome to stimulate IgA broadly to the entire microbiome as occurs with pectin derivative treated mice. The investigator's goal will be to isolate the microbes that respond to fiber to alter levels of IgA in the gut lumen.

DETAILED DESCRIPTION:
Participants will be either selected from a pool of previously screened and identified candidates or who have communicated interest in participating in research through GoodNature Program, run by Aimmune. No participants who have made or have potential to make a lot of a finished product will be allowed to participate. Those who agree to participate will complete a health pre-screening survey over electronic form or phone call and complete the informed consent form (ICF). After completion of the ICF, participants will be assigned a unique, anonymous participant ID. Only a select few members of the Study Sponsor will have access to the identification codes; deidentification codes will not be shared with collaborators. Following this, participants will be given general information regarding diet practices, fiber benefits, and details regarding the study, including sample collection and labeling of samples, diet tracking via surveys, photos of meal submissions, etc.

Participants will meet at a study site and will be provided with chia seeds, the manual stool sampling tool, and pre-labeled specimen containers if they are collecting their samples at home. At this time, participants may also provide blood specimens.

Once the pre-intervention materials are completed, participants (60) will begin a 16-week intervention period; half of participants will add daily 2.5 tbsp chia seeds for the first 8-weeks of the study and return to their normal diet for the second 8-weeks, half of participants will maintain their normal diet for the first 8-weeks and add daily 2.5 tbsp chia seeds for the second 8-weeks as a crossover design. Multiple people in the household can participate, but because we want to understand transmissibility of SCFU and/or IgA levels.

Participants will be randomized into two groups, but members of the same household will be assigned into opposite groups.

All participants will be asked to complete a short, electronic daily stress survey, including providing daily photos of meals. The daily survey will include the Patient Health Questionnaire (PHQ-4), a brief validated screening questionnaire consisting of a 2-item depression scale (PHQ-2) and a 2-item anxiety scale (GAD-2)2. The PHQ-4 data will be used to track stress. Daily photos of meals will be used to track diet data throughout the study.

PHQ-4 total score ranges from 0 to 12, with categories of psychological distress being2:

* None 0-2
* Mild 3-5
* Moderate 6-8
* Severe 9-12

Anxiety subscale = sum of items 2 and 3 on Daily Survey Form (score range 0 to 6) Depression subscale = sum of items 4 and 5 on Daily Survey Form (score range 0 to 6) On each subscale, a score of 3 or greater is considered positive for screening purposes.

Participants will be also be asked to collect a minimum of 3 stool samples per week during the study. Participants who are collecting stool samples at home will store samples in their freezers in a provided biohazard storage container and samples will be picked up weekly by study staff or a courier. All participants will scan the QR code on the container to record the sample collection date and time and will write the collection date on the container.

On weeks 1, 8, and 16, participants will be asked to collect detailed diet data via electronic survey, using the NIH Automated Self-Administered 24-Hour Dietary Assessment Tool. Stool samples will be prepared and aliquoted by the Study Sponsor and sent to UCI and Cleveland Clinic for bacterial PCR, Metabolomic analysis, Shotgun metagenomic sequencing, bacterial spore titer evaluation, and IgA Testing. All samples, including blood samples, will be retained indefinitely in a -80C freezer at Aimmune Therapeutics for research per the existing Biobank Protocol #20234092. Mid- and post- intervention surveys will be sent to participants to evaluate experiences with the study and chia seeds, as well as to identify any side effects or complaints.

Deidentified surveys will be provided to and analyzed by the Study Sponsor.

IgA low subjects throughout the study. To discover the unknown IgA-degrading bacteria, researchers will spread fecal samples of IgA-Low subjects on CDC anaerobic blood agar plates to form single colonies. Next, researchers will subculture all the colonies on new CDC blood agar by streaking. Researchers will scrape each subculture colony into sterile PBS buffer and pool ~15 individual colonies for the in vitro incubation with IgA and Pigr. After overnight incubation at 37 °C, WB analysis will be used for evaluation of the degradation of IgA and Pigr. Colonies from the bacterial pool with IgA/Pigr-cleaving activity will be individually incubated with the substrates again and analyzed by immunoblotting.

Evaluate complexity of IgA degrading bacteria. Researchers will determine antibiotic sensitivities of the candidate bacteria in vitro. Because of the challenges with T. immunophilia (IgA degrader in mice), researchers will evaluate the complexity of colonies (are they easily grown in pure culture versus the presence of companion bacteria within the isolated colony). If the candidate IgA degrader grows slowly in culture, researchers will evaluate the bacteria for auxotrophy as for T. immunophila. Researchers will use genomic and metabolic tools in combination to test for auxotrophy.

IgA high subjects at the end of the study. Researchers will inoculate germ free mice with stool samples from these donors and evaluate IgA levels after two weeks in these mice (we will IgA low samples as a control). For mice that have high levels of IgA, researchers will isolate spores be various methods and test in germ free mice. Researchers will refine the IgA stimulating community as much as is possible and test if it is culturable. The goal is to identify human gut microbes that respond to fiber in the diet and alter IgA levels to all gut microbes.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or greater
2. Able to sign informed consent in English
3. Households (2 or more adults) or individuals who are willing to provide a minimum of 3 separate stool samples per week and utilize a manual stool sampling tool. Alternatively, participants who can come to a collection site and leave stool samples a minimum of 3 days per week throughout the duration of the study.
4. Are generally healthy
5. Agreeable to adding chia seeds to diet
6. Have access to a smartphone

Exclusion Criteria:

1. Less than 18 years of age
2. Greater than 50 years of age
3. Unable to provide a minimum of 3 stool samples per week
4. Active donors for a commercial product
5. Anyone who previously made a lot of a finished product
6. Diagnosed with a digestive, intestinal, or other condition that contraindicates consuming a daily serving size of chia seeds (~2.5 tbsp).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Stool SCFU (Spore Colony-Forming Units) | 8 weeks
  Evaluate the impact of increased dietary fiber (an estimated additional 10 g per day) on stool SCFU (Spore Colony-Forming Units).

SECONDARY OUTCOMES:
Stool SCFU (Spore Colony-Forming Units) | 16 weeks
  Evaluate the effect of stress on stool SCFU in biological samples collected from healthy donors
Biomarkers and Microbiome Composition | 16 weeks
  Stool Bacterial spore titers will be compared against stool whole metagenomic sequencing results and stool IgA results to determine any correlations between these variables.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Goldsmith, MD, PhD, Principal Investigator — Nestle Health Science
Locations (2):
- United States (2):
  - Aimmune Therapeutics Manufacturing, Ambler, Pennsylvania
  - GoodNature Tempe, Ambler, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Beginning 6 months and ending 2 years after the publication of results
Access Criteria: Proposals must be submitted to the Sponsor to receive the IPD and data analysis through a commercially available portal. The URL is not currently available but will be made available after the study is published.